CLINICAL TRIAL: NCT05086107
Title: An Open-label, Non-randomized, Monocenter, Single-dose, Phase I Study to Evaluate Pharmacokinetics and Safety of BV100 Administered as Single Intravenous In-fusion to Subjects With Renal Impairment
Brief Title: Pharmacokinetics and Safety of BV100 Administered as Single Intravenous Infusion to Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Collaborators: Clinical Research Units Hungary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: BV100-003
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-06

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Rifabutin

STUDY DESIGN:
Intervention Model Description: BV100 administered as a single intravenous infusion to subjects with varying degree of renal impairment and control volunteers with normal renal function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): subjects with mild renal impairment (eGFR: 60 to 89 mL/min)
  Interventions: Drug: BV100
- Group 2 (Experimental): subjects with moderate renal impairment (eGFRr: 30 to 59 mL/min)
  Interventions: Drug: BV100
- Group 3 (Experimental): subjects with severe renal impairment (eGFR: 15-29 mL/min)
  Interventions: Drug: BV100
- Group 4 (Experimental): subjects with normal renal function (eGFR: ≥ 90 mL/min)
  Interventions: Drug: BV100
- Group 5 (Experimental): subjects with end stage renal disease (ESRD) eGFR: <15 mL/min requiring dialysis (with BV100 dosing and PK during the dialysis-free interval)
  Interventions: Drug: BV100
- Group 6 (Experimental): subjects with ESRD (eGFRr: <15 mL/min) requiring dialysis (with BV100 dosing and PK on the day of dialysis)
  Interventions: Drug: BV100

INTERVENTIONS:
Drug: BV100 — Rifabutin for infusion
  Other Names: Rifabutin for Infusion

SUMMARY:
To investigate the pharmacokinetics (PK) of rifabutin in subjects with renal impairment after single intravenous (IV) infusion of BV100

DETAILED DESCRIPTION:
To investigate the pharmacokinetics (PK) of rifabutin and excipient in subjects with renal impairment after single intravenous (IV) infusion of BV10=. In addition to investigate the safety and tolerability of BV100 in subjects with renal impairment and to investigate the PK of 25-acyl-rifabutin metabolite in subjects with renal impairment after single intravenous (IV) infusion of BV100

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and follow instructions during the study.
2. Subjects who signed informed consent.
3. Male subjects ≥18 and ≤75 years of age; female subjects ≥18 and ≤75 years of age of non-childbearing potential, defined as follows:

   * female subjects 50 years of age or older, in menopause for 24 consecutive months, and not receiving any hormone replacement therapy within 24 months prior to inclusion into the study
   * female subjects who underwent surgical sterilization
   * female subjects who underwent hysterectomy
   * female subjects with documented premature ovarian failure
4. Weight within a BMI range of 19.0-35.0 kg/m2, range limits inclusive.
5. Having had no febrile or infectious illness for at least 7 days prior to dosing.
6. The subject will be available to complete the study.
7. The subject commits to comply with the restrictions and requirements of the protocol and, in the opinion of the study physician, will be able to complete the study.

   Control volunteers with normal renal function, in addition to criteria of "All subjects":
8. Estimated glomerular filtration rate (eGFR) according to MDRD:

   * ≥90 mL/min (normal renal function)
9. Control subjects have to be in good health or in stable condition, in the opin-ion of the study physician, as determined by medical history, ECG, vital signs, physical examination, and clinical laboratory tests. Subjects having chronic conditions should have an onset of at least 3 months prior to Screening, clini-cally stable, and well-controlled.

   Renally impaired patient volunteers, in addition to criteria of "All subjects":
10. Estimated glomerular filtration rate (eGFR) according to MDRD:

    * 60-89 mL/min (mild renal impairment)
    * 30-59 mL/min (moderate renal impairment)
    * 15-29 mL/min (severe renal impairment)
    * <15 mL/min (requiring dialysis)
11. Stable renal impairment, defined as no clinically significant change in dis-ease status within 2 weeks from Screening, as judged by the Investigator.
12. Subjects with systolic blood pressure ≥ 90 mmHg and diastolic blood pressure ≥ 50 mmHg.
13. Patients with chronic diseases / conditions other than renal impairment can be included, provided that these diseases / conditions are stable, well-controlled, and do not interfere with the study objectives or the subject's over-all safety, as judged by the Investigator.

Exclusion Criteria:

1. Unwilling or unable to give informed consent.
2. As a result of the medical screening process, the study physician considered the subject unfit for the study.
3. Pregnant or lactating women or men with female partners who are lactating or are pregnant.
4. Known or suspected history of hypersensitivity to rifabutin or excipients or to drugs of a similar chemical class including rifampicin, rifapentine, rifaximin; history of allergic reactions leading to hospitalisation or any other allergic con-ditions (including drug allergies, asthma, eczema, anaphylactic reactions but excluding untreated, asymptomatic, seasonal allergies) which the Investigator considers may affect the safety of the subject and / or the outcome of the study.
5. History of antibiotic-associated diarrhoea within one year.
6. Subjects with significant ECG abnormalities (history, or evidence of sec-ond-degree heart block of Mobitz type II, third degree heart block, or any ab-normality considered relevant by the Investigator), QTcF > 460 ms, PR > 200 ms, or QRS duration > 120 ms.
7. History of symptomatic, chronic or recurrent infection (e.g. nausea, vomit-ing, diarrhoea, infection with fever) or any viral, bacterial, fungal or parasitic infection within 30 days prior to admission to the clinical unit.
8. A positive screening serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)-1 and / or 2.
9. Positive drugs-of-abuse or alcohol screen.
10. History of epilepsy, other neurological disorders, or neuropsychiatric con-ditions.
11. History of seizures.
12. Subjects having used megadose vitamins (i.e. 20 to 600 times the recom-mended daily supplement dose) within 7 days prior to dosing, unless in the opinion of the study physician the medication does not interfere with the study procedures or compromise safety
13. Volunteers who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes, utilized within 30 days of IMP administration.
14. Regular use within 3 months of IMP administration of a CYP3A enzyme modifier - any inhibitor, moderate or strong inducer, and sensitive or moder-ately sensitive substrate, as listed in Section 11.3 'Prohibited concomitant med-ications'.
15. Volunteers who have participated in a clinical study involving administra-tion of an investigational drug within the following time period prior to the dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
16. Volunteers who consume more than 21 units of alcohol per week, or who have a significant history of alcohol abuse (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 30 mL of 40% of alcohol by volume distilled spirits).
17. Excessive consumption of caffeine- or xanthine-containing food or bever-ages (> 5 cups of coffee a day or equivalent), or inability to stop consuming from 48 hours prior to study treatment administration.
18. Subjects who smoke more than 10 cigarettes a day.
19. Any use of drugs-of-abuse or alcohol abuse within 2 years prior to the first admission to the clinical unit.
20. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the requirements of the study.
21. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct. Failure to satisfy the Investigator of fitness to participate for any other reason.
22. Any significant blood loss, donation of one unit (450 mL) of blood or more, or receipt of transfusion of any blood or blood products within 60 days, or plasma donation within 7 days prior to the first admission to the clinical study site.
23. Volunteers who are employees or immediate family members of the study site or Sponsor.

    Control volunteers with normal renal function, in addition to criteria of "All subjects":
24. Supine systolic blood pressure > 150 mmHg or < 90 mmHg, or diastolic blood pressure > 100 mmHg or < 50 mmHg at Screening or on Day 1, prior to dosing (any abnormal blood pressure results may be repeated arbitrarily, and if the repeat result is within the normal range, it is not considered to have met the exclusion criterion). Pulse rate > 100 or < 50 beats per minute at Screening or on Day 1, prior to dosing.
25. Screening laboratory values should not exceed 1.5 x ULN, and the eventu-al deviation should be deemed as being clinically non-significant. Any abnor-mal value of these parameters may be repeated arbitrarily, and if the repeated result is within the allowed range, it is not considered to have met the exclusion criterion.
26. Volunteers who have received any new prescribed systemic or topical medication within 4 weeks of the first dose administration.

    Renally impaired patient volunteers, in addition to criteria of "All subjects":
27. Acute renal failure (as judged by the Investigator).
28. History of kidney transplant regardless of functionality.
29. History of nephrectomy.
30. Start of any new medication or any changes to current dosages within 14 days prior to study drug administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
To investigate the pharmacokinetics (PK) of rifabutin in subjects with renal impairment | 96 hours
  Area under the plasma concentration versus time curve (AUC)
To characterize the single dose pharmacokinetic profile of rifabutin | 96 hours
  Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
To investigate the safety and tolerability of single intravenous ascending doses of BV100 assessed by the nature, occurrence, and severity of treatment-emergent adverse events | 7 days
  Safety and Tolerability
To determine the plasma concentration of the main metabolite 25-O-Desacetyl-Rifabutin in plasma in subjects with renal impairment | 96 hours
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- CRU Hungary Kft., Early Phase Unit, Miskolc, Hungary

IPD SHARING:
Plan to Share IPD: No